CLINICAL TRIAL: NCT06311474
Title: Assessment and Treatment of Behavior Problems in TSC at Preschool Age: A Telehealth Approach
Brief Title: Remote Assessment and Intervention for Behavior Problems in Kids With TSC
Acronym: RAINBOW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nicole McDonald, PhD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-22-1-0250
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Tuberous Sclerosis
Keywords: TAND; TSC; Behavior Problems; PCIT; TSC-Associated Neuropsychiatric Disorders
MeSH Terms: conditions — Tuberous Sclerosis; Mental Disorders

STUDY DESIGN:
Intervention Model Description: The clinical trial portion of this study uses a waitlist control design with random assignment to group. Randomization is stratified by age (3-4 years old, 5-6 years old).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by assessors who are blind to group status. Investigators will be kept blind to study outcomes until data collection for the primary outcome is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control (No Intervention): Participants randomized to the waitlist control (or delayed treatment) condition will receive written and verbal feedback after the baseline assessment visit. These families will participate in follow-up visits at 3 months, 6 months, and 12 months after the baseline visit. They will receive the same treatment (PCIT) after the 6-month assessment.
- Immediate Treatment (Experimental): Participants randomized to the immediate treatment condition will receive written and verbal feedback after the baseline assessment visit. These families will begin PCIT shortly after this visit. These families will participate in follow-up visits at 3 and 6 months after the baseline visit.
  Interventions: Behavioral: Parent-Child Interaction Therapy (PCIT)

INTERVENTIONS:
Behavioral: Parent-Child Interaction Therapy (PCIT) — PCIT is a dyadic therapy that focuses on enhancing the parent-child relationship and improving child behavior through positive parenting and limit setting skills. All PCIT sessions are delivered remotely via Zoom once per week for up to 20 weeks. Session length is about 1 hour. There are two distinct phases of PCIT, the Child Directed Interaction and the Parent Directed Interaction. Each phase begins with a Teach session, where parents learn about the skills they will practice during that portion of PCIT, and is followed by Coach sessions, in which the PCIT therapist provides direct feedback and live coaching on the use of the skills. An additional component is Daily Play practice. Parents are instructed to spend five minutes per day playing with their child, during which they practice skills learned during sessions. Adaptations have been made to the standard approach to increase suitability for the TSC population.
  Arms: Immediate Treatment

SUMMARY:
The RAINBOW study is a fully remote study focused on understanding and treating behavior problems in young children with tuberous sclerosis complex (TSC). The first goal is to enroll a group of 100 children with TSC between the ages of 3 and 6 years old, with and without problem behaviors, to learn about how best to measure behavioral challenges in TSC and how common these behaviors are during this age period. All families will get feedback from the clinical assessments collected. Eligible children who are experiencing behavior problems will be invited to enroll in a pilot clinical trial of internet-based Parent-Child Interaction Therapy (or PCIT), which is meant to help parents better manage their children's challenging behaviors. Adaptations to PCIT are incorporated to suit the needs of TSC children and families. Some participants will be randomly selected to receive the intervention immediately and others after a 6-month delay, but all families will receive the same intervention. Intervention sessions occur on a weekly basis for up to 20 weeks. Follow-up assessments, which include play interactions, parent interviews, and questionnaires occur about 3 and 6 months after the first visit. The delayed treatment group has an extra brief assessment about 12 months from the initial visit. This study will increase what is known about the types of behavior problems that come up during preschool age in TSC and how best to help children and families with TSC who are experiencing these problems.

DETAILED DESCRIPTION:
The proposed study uses a telehealth approach to remotely assess and treat behavior problems in preschool-aged children with TSC. This study aims to 1) measure the prevalence and quality of externalizing behavior problems and their relation to family functioning in preschool-aged children with TSC; 2) examine the feasibility and acceptability of internet-based PCIT (I-PCIT) in children with TSC; 3) investigate the effects of I-PCIT on child and parent behavior in preschool-aged children with TSC and behavior problems; and 4) examine predictors of treatment response.

For Aim 1, 100 children with TSC ages 3-6 years old will be enrolled. Developmental abilities and behavior problems will be assessed using norm-referenced parent report measures and video recordings of parent-child interactions. The prevalence of behavior problems in young children with TSC and relation to family functioning will be assessed. A subset of the children from Aim 1 who exhibit elevated externalizing behavior will be recruited for the pilot intervention, with a target sample size of 32. Children will be randomized to an immediate treatment or waitlist control group. Assessments will be performed at baseline (using Aim 1 data), mid-point (3 months later), and post-treatment (6 months later). Families randomized to the waitlist group will have a brief, additional post-treatment assessment 12 months post-baseline). Sessions occur on a weekly basis for up to 20 weeks. Preliminary efficacy will be examined by comparing trajectories from baseline to post-treatment between the immediate treatment and waitlist control groups. Data on feasibility, acceptability, and predictors of treatment response will be studied across all intervention participants.

ELIGIBILITY:
Inclusion Criteria:

For assessment visit:

* Clinical diagnosis of TSC
* Chronological age of 3 years, 0 months to 6 years, 11 months old at enrollment.
* English or Spanish as primary language in the home.

For intervention study only:

* Elevated behavior problems
* Parent/caregiver available to participate in PCIT

Exclusion Criteria:

For assessment visit:

* None

For intervention study:

* Plan for epilepsy surgery during study period

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory (ECBI) | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up (delayed treatment group only)
  The ECBI is a norm-referenced caregiver report measure of disruptive behavior in children.

SECONDARY OUTCOMES:
Behavior Assessment Scale for Children-3rd Edition (BASC-3) | Baseline, 6-month follow-up
  The BASC-3 is a norm-referenced caregiver report measure of broad behavior problems and adaptive skills in children.
Vineland Adaptive Behavior Scales-3rd Edition (Vineland-3) | Baseline, 6-month follow-up
  The Vineland-3 is a norm-referenced caregiver report measure of adaptive skills for infancy through adulthood. Communication, daily living, socialization, and motor skills are measured. The parent interview version is used for this study.
Parenting Stress Index-4th Edition-Short Form (PSI-4-SF) | Baseline, 6-month follow-up
  The PSI-4-SF is a norm-referenced self-report measure of parenting-related stress.
Dyadic Parent-Child Interaction Coding System (DPICS) | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up (delayed treatment group only)
  The DPICS measures parent-child interactions across 3 situations: child led play, parent led play, and clean up. Language and behavior are coded according to the DPICS-IV coding system.
Therapy Attitude Index (TAI) | 6-month follow-up (immediate treatment), 12-month follow-up (delayed treatment)
  The TAI measures treatment acceptability in PCIT.
Telehealth Usability Questionnaire (TUQ) | Baseline & 6-month follow-up (immediate treatment), 6-month follow-up & 12-month follow-up (delayed treatment)
  The TUQ measures comfort with the use of telehealth methods pre- and post-treatment.
Aberrant Behavior Checklist (ABC) | Baseline, 6-month follow-up
  The ABC is a caregiver report questionnaire commonly used to measure problem behaviors and behavior change in children and adults with disabilities.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole McDonald, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided